CLINICAL TRIAL: NCT06416917
Title: Prevalence of Glenohumeral Internal Rotation Deficit Among Selected Professional Athletes
Brief Title: Glenohumeral Internal Rotation Deficit Among Professional Athletes
Status: Recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hadeel Ibrahim Ali, assistant lecturer, Cairo University
Other Study IDs: prevalence of GIRD
Record Dates: First submitted 2024-05-12; First posted 2024-05-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Internal Rotation Contracture-shoulder
Keywords: GIRD

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: bubble inclinometer — to measure range of motion

SUMMARY:
The study aimed to identify the prevalence of GIRD among elite Egyptian volleyball players in selected clubs in Egypt.

DETAILED DESCRIPTION:
Volleyball is a highly technical sport that involves powerful overhead movements performed repetitively. The volleyball attack "spike," is a complex overhead movement that professional players perform up to 40,000 times a year (Kugler, 1996). It consists of four phases: windup, cocking, acceleration, and deceleration (follow-through). The windup phase is the arm is elevated to a position that is more than 90° from the anatomical position and the shoulder is slightly horizontally abducted. The cocking phase is abduction and external rotation (ER) reach their maximum levels. The acceleration phase is the shoulder rapidly internally rotates and adducts the arm up to the point where the hand strikes the ball (shoulder abducted at 140°-170° in neutral rotation. The deceleration (follow-through) phase extend from ball impact until the arm finally stops on the side of the trunk (Seminati et al., 2015).

The shoulder complex has the widest multi-planar range of motion (ROM), it is a frequently injured body part in volleyball (12%-18%), mainly due to overuse mechanisms (Agel et al., 2007; Clarsen et al., 2015; Cuñado-González et al., 2019). Shoulder injuries are the third-most common volleyball injury (Reeser et al., 2010), According to reports, between (15- 23%) of volleyball players experience shoulder pain or injuries during a season (Clarsen et al., 2015; Cuñado-González et al., 2019; Forthomme et al., 2013). As a result, shoulder injuries are the most common reason for missing volleyball matches and practices (Hao et al., 2019).

Glenohumeral internal rotation deficit (GIRD) is an adaptive process in which the throwing shoulder has a loss of internal rotation (IR) ROM (Rose & Noonan, 2018). The anatomical GIRD is a typical response in overhead athletes with a lowered IR of about 18̊ to 20⁰ and symmetry in the total rotation motion (TRM), while Pathologic GIRD was identified in athletes with an IR deficit greater than 18⁰ and a TRM difference of more than 5⁰ between the shoulders. Not all cases of GIRD are indicative of pathology (Manske et al., 2013).

It has been reported that GIRD can be seen in athletes who play softball, tennis, handball, football, baseball and even javelin throwers (Mlynarek & Lee, 2017). Most of the studies are involved in baseball players, while volleyball and other overhead sports are known to have different throwing kinematics (Reeser et al., 2010). It has been shown that asymptomatic overhead athletes have GIRD at 10-15° whereas symptomatic overhead athletes have GIRD at 19-25° (Kaplan et al., 2011; Myers et al., 2006; Trakis et al., 2008). A higher degree of GIRD was found in the pain group than the no-pain group on symptomatic and asymptomatic handball and tennis players (Almeida et al., 2013; Moreno-Pérez et al., 2015). However, Lubiatowski et al., (2018) found only eleven out of eighty-seven handball players exhibited GIRD, although the author did not account for GIRD unless it reached 20-25°. Ellenbecker et al., (2002) have reported decreases of 5-10 ⁰ on average in the dominant arm TRM parameter in uninjured elite-level tennis players. Regarding volleyball, some authors found that few asymptomatic volleyball players displayed GIRD, but unless a player had a GIRD of > 18°, they did not consider them to have GIRD (Harput et al., 2016; Saccol et al., 2016).

Mizoguchi et al., (2022) studied (123 male and female) of adolescent (15 to 17 years old) volleyball players in Japan and found 38.2% had GIRD and decreased TRM in their shoulders. The GIRD group had an intrinsic external rotation deficiency (ERD) that was unrelated to sex, body composition, a history of shoulder injuries, years of volleyball experience, practice time, or court position. There were sex-specific differences in shoulder ROM, especially in the external rotation (ER) and IR ROM, with males being hypomobile and females being hypermobile. These results find agreement with (Harput et al., 2016) who found that 38.5% of adolescent volleyball players had GIRD with decreased TRM. Reeser et al., (2010) discovered a significant GIRD (8.9°), a non-significant presence of external rotation gain (ERG) (2°), and no change in TRM. It was reported in literature that There is still much to learn about the connection between volleyball players' shoulder pain and GIRD, so more research is required (Schmalzl et al., 2022; Harput et al., 2016).

It was found that GIRD is often present in adult volleyball players (Schmalzl et al., 2022), but this may not be related to shoulder pain or injury, but imbalances in muscle strength around the shoulder can affect pain or injury (challoumas et al., 2017). The offensive players of volleyball players have a GIRD of ≥10 ⁰ and a lower TRM are linked to a higher prevalence of posterior-superior impingement (Schmalzl et al., 2022).

Alqarni et al., (2022) showed that GIRD was present in pain group and no pain group. The pain group exhibited higher degrees of GIRD (15.65°) than the no pain group (9.06°). The results also revealed that the pain group exhibited a higher difference in TRM (16.17°) than the no pain group (10.17°).

Players of volleyball may have changes in glenohumeral (GH) joint mobility and flexibility as a result of their sport-related activities (Harput et al., 2016; Keller et al., 2018; Wilk et al., 2011; Burkhart et al., 2003). They commonly perform spiking and serving (Reeser et al., 2010), which causes the shoulder joint to modify its bony and soft tissue structures. This results in 8-20% of all volleyball players' injuries (Reeser et al., 2010). Deceleration might result in repeated microtrauma as a consequence of the alteration in shoulder biomechanics during throwing exercises. This adaptation is essential for performance, yet it can also be a risk factor for injuries, leading to questions about how much of this deficit can be tolerated before clinical intervention is required (Whiteley & Oceguera, 2016).

In summary, GIRD is a common condition in volleyball players. It is not always associated with pain or injury, but it can be a risk factor for posterior-superior impingement. Up to author knowledge, there is no published study regarding the prevalence of GIRD among professional Egyptian volleyball players.

ELIGIBILITY:
Inclusion Criteria:

* 1. A professional volleyball Egyptian athlete who are playing in the selected clubs around Egypt; the four clubs in Alexandria (Smouha sporting club, Alex sporting club, Ittihad club and Horse owners club) and the three clubs in Cairo (Egyptian shooting club, wadi degla club, Zamalek club).

  2. Elite Male and female volleyball players with BMI between (18.5 to 24.9) kg/m².

  3. Their age range is between 14 to 30 years old

Exclusion Criteria:

* 1. Athletes who have a history of shoulder surgery or injury such as rotator cuff tear or labrum tear.

  2. Athletes who have a history of injuries (fractures, dislocations) or surgeries in other joints of the upper limb (elbow, forearm, wrist, and hand) (Dabhokar et al., 2018).

  3. Athletes who have a history of inflammatory joint disease, or neurological disorders that could affect their shoulder ROM such as arthritis or diabetes (Dabhokar et al., 2018).

  4. Athletes who are taking any medications that could affect their shoulder ROM or pain.

  5. Athletes who are currently inactive at the professional level due to multiple injuries that have prevented them from practicing.

  6. Athletes who have been diagnosed with kyphosis and scoliosis in the shoulder and thoracic regions, as well as other anatomical anomalies (pennella et al., 2022).

  7. Athletes who have experienced shoulder pain with stomach discomfort (pennella et al., 2022)

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: professional volleyball athletes from 18 to 30 years old.
Sampling Method: Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2024-09-29 (Estimated); Study Completion 2024-10-30 (Estimated)

PRIMARY OUTCOMES:
internal rotation, external rotation and total range of motion | 4 months
  shoulder range of motion
physical performance | 4 months
  questionnaire
pain intensity | 4 months
  visual analog scale

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Physical Therapy, Cairo, Egypt